CLINICAL TRIAL: NCT04523948
Title: Comparative Tobacco Interventions for Individuals With Severe and Persisting Behavioral Health Disorders
Acronym: THRRP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Sponsor
Other Study IDs: GG-0037
Record Dates: First submitted 2020-07-23; First posted 2020-08-24 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Tobacco Use
Keywords: Mental Heatlh; Substance Use; Harm Reduction
MeSH Terms: conditions — Tobacco Use; Substance-Related Disorders; Harm Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort One: Subjects will be invited to participate in brief weekly in person or telehealth behavioral support with the objective of reducing their rate of combustible tobacco use. Subjects will also be offered the choice of various conventional nicotine replacement aids, snus, electronic cigarette, varenicline or bupropion.
  Interventions: Behavioral: Behavioral and pharmacological support to reduce combustible tobacco use.
- Cohort Two: Subjects will be invited to participate in brief weekly in person or telehealth behavioral support with the objective of reducing their rate of combustible tobacco use. Subjects will also be offered the choice of various conventional nicotine replacement aids, snus, electronic cigarette, varenicline or bupropion.
  Interventions: Behavioral: Behavioral and pharmacological support to reduce combustible tobacco use.
- Cohort Three: Subjects will be invited to participate in brief weekly in person or telehealth behavioral support with the objective of reducing their rate of combustible tobacco use. Subjects will also be offered the choice of various conventional nicotine replacement aids, snus, electronic cigarette, varenicline or bupropion.
  Interventions: Behavioral: Behavioral and pharmacological support to reduce combustible tobacco use.
- Cohort Four: Subjects will be invited to participate in brief weekly in person or telehealth behavioral support with the objective of reducing their rate of combustible tobacco use. Subjects will also be offered the choice of various conventional nicotine replacement aids, snus, electronic cigarette, varenicline or bupropion.
  Interventions: Behavioral: Behavioral and pharmacological support to reduce combustible tobacco use.
- Cohort Five: Subjects will be invited to participate in brief weekly in person or telehealth behavioral support with the objective of reducing their rate of combustible tobacco use. Subjects will also be offered the choice of various conventional nicotine replacement aids, snus, electronic cigarette, varenicline or bupropion.
  Interventions: Behavioral: Behavioral and pharmacological support to reduce combustible tobacco use.

INTERVENTIONS:
Behavioral: Behavioral and pharmacological support to reduce combustible tobacco use. — Behavioral and pharmacological support to reduce combustible tobacco use.

SUMMARY:
The aim of this pilot intervention is to examine the acceptability of a harm reduction intervention approach to tobacco use for individuals with serious behavioral health disorders and its association with a decrease in smoking. The intervention uses a "dynamic" approach to patient choice, allowing participants the option to explore different strategies for harm reduction, while providing support from counselors in the process. Therefore, the investigators have chosen an observational study design in order to document and explore the acceptability and outcomes of the intervention.

DETAILED DESCRIPTION:
Background and Significance

The high rate of combustible tobacco use among persons with schizophrenia, affective, post traumatic stress and substance misuse disorders is well documented. Over 40% of the estimated 9.8 million Americans, or 4.0% of the total population, who have serious behavioral health disorders smoke cigarettes, at a rate two to three times higher than the general population. The adverse health consequences and abbreviated lifespan for these persons is also well documented. Given the greater rate of tobacco use, persons with behavioral health disorders are at greater risk for morbidity, e.g., respiratory and cardio-vascular illness, and pre-mature mortality. The relationship of individuals in these communities to combustible tobacco in its pharmacological, sensorimotor and behavioral aspects is compelling. There is a significant literature documenting the endorsement and benefit of nicotine and smoking behavior for individuals in these communities.

Clinical or personal context contribute to the barriers in making change, e.g., the social acceptability of smoking, lack of support, poor access to interventions, the need to mitigate stress and other symptoms of serious mental illness. The need for meaningful structure and daily engagement leads many to use tobacco to fill time and as a distraction. However, many individuals express a desire to quit or further reduce their tobacco consumption. Conventional tobacco interventions and approaches, e.g., smoking cessation, quit lines, informal telephone counseling, FDA approved Nicotine Replacement Therapies (NRTs) and medications have limited documented success. Existing evidence indicates that the combination of pharmacological intervention along with behavioral support is superior to either of these interventions alone. However the behavioral support aspect is usually limited to four to eight sessions.

Local Need

As documented by the State,California has led the way in the progressive decrease in combustible tobacco use. San Francisco County has a 10.8% rate of smoking. Over 25,000 adults received service on an annual basis from the San Francisco Department of Public Health. Of these service recipients at least 6028 adults or 24% (18 or older) are smokers, 5722 persons report having never smoked and for another 7926 (31.5%) smoking status is unknown. The larger department of public health offers smoking cessation services however there are no dedicated services targeting the behavioral health service user. Tobacco use is increasingly of concern for behavioral health program administrators and managers. Recruitment of programs for this research effort was met with enthusiasm and an unambiguous expression of a need for an intensive, harm reduction approach to tobacco intervention. The local Health Department division of Behavioral Health Services maintains a dedicated Harm Reduction policy regarding substance use behaviors.

Consultants were retained to conduct, record and analyze the experience, barriers, challenges and satisfaction with smoking and smoking cessation attempts for individuals with behavioral health disorders through the facilitation of four focus groups. In summary, focus group participants report an understanding of smoking as an addiction integral to their daily lives; that its pleasurable effects override health concerns; that cigarettes are a "friend" and something to pass time and overcome boredom; that they understood restrictions on smoking but also feel harassed or demeaned for smoking; and that not smoking requires "willpower" against a powerful addiction. Some felt that a "harm reduction" approach, e.g., gradual reduction was best and most acknowledge that relapse was a common experience. There was a wealth of experience with smoking cessation and a diversity of satisfaction with various intervention strategies. Gum and patch were generally reported as not satisfying; Chantix was found to be helpful and a curiosity about inhaler or vaping as long as it is safe. Individuals also reported on personal strategies to help with reduction or cessation. More generally, individuals wanted more information about the range of choices. Some noted that access through insurance was a barrier except for those who had both Medicaid and Medicare. It is notable that participants report that they did not appreciate preaching or lecturing about the need to stop smoking. The conclusion is that individuals express a desire to reduce or abstain from tobacco use and also express the need for more help in doing so. Interest in the various intervention choices is diverse however gradual reduction with some aide appears to be the modal choice.

Hypotheses

1. A Harm Reduction approach will result in a decrease in daily combustible tobacco use when compared to baseline use.
2. Support and harm reduction approaches will be important to acceptability.

Research Questions

1. Does this Harm Reduction approach reduce combustible tobacco use when compared to baseline use?
2. Which strategies or combination of strategies demonstrate a greater or lesser impact in combustible tobacco use?
3. At what service intensity points, e.g., intervention dose as defined by number of weeks, does combustible tobacco use decrease?
4. To what degree does this Harm Reduction approach retain individuals in this intervention, i.e., acceptability of intervention?
5. What are participants' experiences with factors that enable success or barriers?

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are formerly or currently being served by San Francisco Bay Area Public Health behavioral health providers. These will include individuals with psychotic, affective, anxiety, personality and substance use disorders.
* Individuals who are not currently enrolled in another formal tobacco intervention or research study.
* Are at least 21 years of age and able to speak English*
* Who score in the "low to moderate dependence" range on the Fagerstrom Test of Nicotine Dependence
* Have used tobacco for at least two years
* Express willingness to participate at least weekly in the intervention strategy
* Express a desire to make some change in their tobacco use pattern
* Express some reason to change their tobacco use pattern
* Have the cognitive capacity to be able to sign a consent to participate in the research

  * A concerted effort will be made to recruit bilingual Chinese and Spanish language staff

Exclusion Criteria:

* The individual does not currently smoke tobacco
* Individuals younger than 21 years of age at the time of enrollment
* Who score in the "low" range on the Fagerstrom Test of Nicotine Dependence
* Have used tobacco for less than two years;
* Express unwillingness to participate at least weekly in the intervention strategy
* Decline an interest in making some change in their tobacco use pattern
* Do not indicate the cognitive capacity to be able to sign a consent to participate in the research

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult individuals who are or have been served by public systems related to a mental health or substance use disorder and are currently using combustible tobacco.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of cigarettes smoked | Change in number of cigarettes smoked per day will be assessed using two time frames: 1) Baseline to 6 months post baseline; and 2) Post intervention which is change from baseline to 12 months post baseline.
  Self-reported number of cigarettes smoked per day
Nicotine Dependence | Change in nicotine dependence will be assessed using two time frames: 1) during the intervention, which is change from baseline to 6 months post baseline; and 2) after the intervention which is change from baseline to 12 months post baseline
  Fagerström Test for Nicotine Dependence, a self-reported scale rated from 0-10, with >=5 indicating dependence (Heatherton et al., 1991).
Carbon Monoxide | Change in carbon monoxide level will be assessed using two time frames: 1) during the intervention, which is change from baseline to 6 months post baseline; and 2) after the intervention which is change from baseline to 12 months post baseline
  Exhaled carbon monoxide level concentration reported in parts per million (ppm) using a breathalyzer assay
Salivary Tobacco Use | Change in salivary nicotine level will be assessed using two time frames: 1) during the intervention, which is change from baseline to 6 months post baseline; and 2) after the intervention which is change from baseline to 12 months post baseline
  Salivary tobacco use level reported in nicotine metabolites (cotinine)

SECONDARY OUTCOMES:
Smoking Decisional Balance | Change in smoking decisional balance will be assessed using two time frames: 1) during the intervention, which is change from baseline to 6 months post baseline; and 2) after the intervention which is change from baseline to 12 months post baseline
  Smoking Decisional Balance is a 6-item self-reported scale which assesses readiness to change in terms of pros (scored from 3-15) and cons (scored from 3-15), based on the Transtheoretical Model of Behavior Change (https://habitslab.umbc.edu/publications/)
Challenges to Smoking Behavior Change | Change in challenges to smoking behavior change will be assessed on two occasions: 1) during the intervention from baseline to 6 months post baseline; and 2) after the intervention which is change from baseline to 12 months post baseline.
  The Challenges to Smoking Behavior Change is a 21 item self-reported scale assessing intrinsic challenges (scored from 9-36) and extrinsic challenges (scored from 12-48) to quitting or reducing smoking (Thomas et al., 2016)
Working Alliance Inventory | Change in working alliance quality will be assessed using two time frames: 1) during the intervention, which is change from baseline to 6 months post baseline; and 2) after the intervention which is change from baseline to 12 months post baseline.
  The Working Alliance Inventory Short Revised version (Busseri & Tyler, 2003) is a 12-item measure that captures three key therapeutic alliance aspects (Horvath & Greenberg, 1989), each scored from 5-20: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond

CONTACTS AND LOCATIONS:
Overall Officials: Kevin McGirr, MS, MPH, Principal Investigator — San Francisco Study Center
Locations (1):
- San Francisco Study Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share IPD.

REFERENCES:
- [Background] Dickerson F, Stallings CR, Origoni AE, Vaughan C, Khushalani S, Schroeder J, Yolken RH. Cigarette smoking among persons with schizophrenia or bipolar disorder in routine clinical settings, 1999-2011. Psychiatr Serv. 2013 Jan;64(1):44-50. doi: 10.1176/appi.ps.201200143. PMID 23280457
- [Background] Evins AE, Cather C, Laffer A. Treatment of tobacco use disorders in smokers with serious mental illness: toward clinical best practices. Harv Rev Psychiatry. 2015 Mar-Apr;23(2):90-8. doi: 10.1097/HRP.0000000000000063. PMID 25747922
- [Background] Glasheen C, Hedden SL, Forman-Hoffman VL, Colpe LJ. Cigarette smoking behaviors among adults with serious mental illness in a nationally representative sample. Ann Epidemiol. 2014 Oct;24(10):776-80. doi: 10.1016/j.annepidem.2014.07.009. Epub 2014 Jul 30. PMID 25169683
- [Background] Hartmann-Boyce J, Chepkin SC, Ye W, Bullen C, Lancaster T. Nicotine replacement therapy versus control for smoking cessation. Cochrane Database Syst Rev. 2018 May 31;5(5):CD000146. doi: 10.1002/14651858.CD000146.pub5. PMID 29852054
- [Background] Jensen AB, Hounsgaard L. "I only smoke when I have nothing to do": a qualitative study on how smoking is part of everyday life in a Greenlandic village. Int J Circumpolar Health. 2013 Aug 5;72. doi: 10.3402/ijch.v72i0.21657. eCollection 2013. PMID 23967409
- [Background] Lindson-Hawley N, Banting M, West R, Michie S, Shinkins B, Aveyard P. Gradual Versus Abrupt Smoking Cessation: A Randomized, Controlled Noninferiority Trial. Ann Intern Med. 2016 May 3;164(9):585-92. doi: 10.7326/M14-2805. Epub 2016 Mar 15. PMID 26975007
- [Background] Lindson-Hawley N, Hartmann-Boyce J, Fanshawe TR, Begh R, Farley A, Lancaster T. Interventions to reduce harm from continued tobacco use. Cochrane Database Syst Rev. 2016 Oct 13;10(10):CD005231. doi: 10.1002/14651858.CD005231.pub3. PMID 27734465
- [Background] Rae J, Pettey D, Aubry T, Stol J. Factors affecting smoking cessation efforts of people with severe mental illness: a qualitative study. J Dual Diagn. 2015;11(1):42-9. doi: 10.1080/15504263.2014.992096. PMID 25491704
- [Background] Schroeder SA, Morris CD. Confronting a neglected epidemic: tobacco cessation for persons with mental illnesses and substance abuse problems. Annu Rev Public Health. 2010;31:297-314 1p following 314. doi: 10.1146/annurev.publhealth.012809.103701. PMID 20001818
- [Background] Stead LF, Koilpillai P, Fanshawe TR, Lancaster T. Combined pharmacotherapy and behavioural interventions for smoking cessation. Cochrane Database Syst Rev. 2016 Mar 24;3(3):CD008286. doi: 10.1002/14651858.CD008286.pub3. PMID 27009521
- [Background] Twyman L, Bonevski B, Paul C, Bryant J. Perceived barriers to smoking cessation in selected vulnerable groups: a systematic review of the qualitative and quantitative literature. BMJ Open. 2014 Dec 22;4(12):e006414. doi: 10.1136/bmjopen-2014-006414. PMID 25534212
- [Background] Uppal N, Shahab L, Britton J, Ratschen E. The forgotten smoker: a qualitative study of attitudes towards smoking, quitting, and tobacco control policies among continuing smokers. BMC Public Health. 2013 May 3;13:432. doi: 10.1186/1471-2458-13-432. PMID 23641875